CLINICAL TRIAL: NCT06764888
Title: Short-Term Outcomes of Minimally Invasive Surgery in Elderly Colorectal Cancer Patients in the Era of ERAS: is a "One-Size-Fits-All" Strategy Sufficient?
Brief Title: ERAS in Elderly Colorectal Cancer Surgery
Acronym: STOMIS-ERAS
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202401646B0
Record Dates: First submitted 2024-12-17; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: ERAS; Colo-rectal Cancer; Elderly (people Aged 65 or More); Minimally Invasive Surgery
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- traditional care group: traditional care group

SUMMARY:
Enhanced recovery protocol consisted of a series of elements aiming to optimize and standardize perioperative care. This study aims to evaluate the safety and feasibility of a modified ERAS protocol following colorectal surgery in the elderly population, aged 65 years or older. This is a retrospective study based on prospectively collected data. Patient privacy has been carefully protected throughout the research process, and no aspect of this study interfered with or altered the patients' treatment or clinical care.

ELIGIBILITY:
Inclusion Criteria:

* they underwent radical resection for colorectal cancer
* the procedure was minimally invasive surgery
* they were aged 65 or older
* they provided signed informed consent.

Exclusion Criteria:

* Patients who underwent emergency surgery for colorectal cancer.
* Patients with incomplete medical records or missing data relevant to the study.
* Patients with synchronous malignancies or a history of other cancers within the past five years.
* Patients with severe comorbidities (e.g., advanced cardiovascular, respiratory, or renal diseases) that contraindicate ERAS protocol implementation.
* Patients with preoperative metastatic disease or locally advanced tumors requiring palliative procedures.
* Patients who did not comply with or complete the ERAS protocol during the perioperative period.

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: From January 2018 to December 2022, comprehensive data on patients who underwent colorectal resection for malignancy at a single medical institute, Chang Gung Memorial Hospital, were prospectively collected and retrospectively reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 1392 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Short-term postoperative complications rate. | 3 months
  Measurement outcomes included the rate of short-term postoperative complications, overall morbidity, early morbidity, reoperation rate, 30-day readmission rates and 30-day mortality rates. Postoperative complications were carefully recorded and classified using the Clavien-Dindo classification system for a standardised severity evaluation. These complications are critical for assessing surgical outcomes and ensuring patient safety. Early complications were defined as those occurring during the initial hospitalisation or within 30 days of surgery, while late complications were defined as those arising after the patient's discharge from the hospital.

SECONDARY OUTCOMES:
Days of Hospital Stay and Time to First Passage of Flatus | 3 months
  Measurement outcomes are the rate of post-operative recovery times, including postoperative stay(days) and first passage of flatus(days).

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided